CLINICAL TRIAL: NCT06013566
Title: SSVEP Evaluation of Brain Function (PRO)
Status: Recruiting | Type: Observational
Sponsor: Headsafe MFG (Industry)
Responsible Party: Sponsor
Other Study IDs: 2018-10-891-PRO
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Mild Traumatic Brain Injury
Keywords: Mild Traumatic brain injury; Concussion; Steady state visual evoked potential; Electroencephalography; Sports Concussion; Sports Medicine
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Baseline: This cohort contains individuals tested at baseline, usually in the pre-season of their sporting season
  Interventions: Device: SSVEP
- Concussed: This cohort contains individuals who have had a concussion, diagnosed by a doctor.
  Interventions: Device: SSVEP
- Suspected Concussion: This cohort contains individuals suspected of having a concussion, but were cleared by a medical professional and do not have a concussion.
  Interventions: Device: SSVEP

INTERVENTIONS:
Device: SSVEP — Non-invasive, non-interventional SSVEP EEG device
  Other Names: Nurochek PRO

SUMMARY:
The investigational device used in this clinical investigation, the Nurochek PRO System (NCPRO), is a portable electroencephalogram (EEG) headset which delivers a visual stimulus and measures a VEP. The visual stimulus is delivered to the subjects' eyes via light-emitting diodes, and the EEG measures the user's visual-evoked potential. This headset communicates with an application on a computer, which processes the signals and transmits them to a secure cloud server for analysis and storage of the data. Nurochek PRO is a development of the previously FDA cleared Nurochek System.

The primary objective of this clinical investigation was to evaluate the performance of the investigational device (NCPRO) against clinical diagnosis of detection of mild traumatic brain injury (mTBI). The primary endpoint outlined for this study was set at the collection of 100 valid investigational device readings from individuals with concussion and 500 valid investigational device readings from healthy individuals who have had a plausible mechanism of sustaining a concussion, but do not have one. Additionally, readings from healthy individuals are also to be acquired.

The aim of this study was to collect data from 100 readings from individuals with concussion. The initial assumption was that sites would provide players pre-season and make players available for testing post-concussion. In practice, some sites provided player data only post-concussion event (such as medical clinics). Participants were acquired from sporting clubs, medical clinicals and schools.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 12 years and older, participating in sport-related activities.

Exclusion Criteria:

* Individuals are excluded if they have a history of seizures, history of epilepsy, structural brain injuries, legal blindness, or sensitivity to flashing lights.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: As above.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Steady State Visual Evoked Potential | 5 days
  A measure of the steady state visual evoked potential (SSVEP) from the device and comparison with a Doctor's diagnosis.

SECONDARY OUTCOMES:
Recovery from m TBI | 30 days
  Follow up testing with the investigational device to examine of there is a link between mTBI recovery and investigational device recordings of brain activity.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Donaldson, MBBS, Principal Investigator — Principal Investigator
Locations (1):
- Headsafe, Sydney, Australia

IPD SHARING:
Plan to Share IPD: No